CLINICAL TRIAL: NCT01313962
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Assessment of the Safety, Tolerability and Pharmacokinetics of Escalating Single Doses of Flufirvitide-3 Nasal Spray in Healthy Subjects
Brief Title: Safety Study of Flufirvitide-3 Nasal Spray in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autoimmune Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIT02-11-01
Record Dates: First submitted 2011-02-16; First posted 2011-03-14 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: antiviral; intranasal; influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flufirvitide-3 (Experimental)
  Interventions: Drug: Flufirvitide-3 0.05 mg single dose; Drug: Flufirvitide-3, 0.1 mg single dose; Drug: Flufirvitide-3, 0.2 mg single dose; Drug: Flufirvitide-3, 0.4 mg single dose
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Flufirvitide-3 0.05 mg single dose — Nasal Spray
  Arms: Flufirvitide-3
Drug: Flufirvitide-3, 0.1 mg single dose — Nasal spray
  Arms: Flufirvitide-3
Drug: Flufirvitide-3, 0.2 mg single dose — nasal spray
  Arms: Flufirvitide-3
Drug: Flufirvitide-3, 0.4 mg single dose — Nasal spray
  Arms: Flufirvitide-3
Other: Placebo — Nasal spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetic profile of flufirvitide-3 nasal spray in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Subjects must be able to understand and be willing to comply with study procedures, restrictions, and requirements.
* Healthy male and non-fertile female subjects aged 18 and 55 years inclusive
* Female subjects must have a negative urine pregnancy test at screening must not be lactating or breastfeeding and must be of non-childbearing potential
* Male subjects should be willing to use barrier contraception during sexual intercourse,
* Body weight 50 to 100 kg inclusive and body mass index (BMI) 18 to 30 kg/m2 inclusive.
* Clinically non-significant findings on physical examination in relation to age.
* Negative Rapid Flu Test (TRU FLU® kit)
* Negative nasal examination upon admission to the study center.

Exclusion Criteria:

* History and/or presence of any clinically significant disease or disorder such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal and psychiatric/mental disease/disorders,
* History and/or presence of hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs. Subjects with a surgical history of the gastrointestinal tract should also be excluded from participation in the study.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the administration of the investigational product which is symptomatic enough to affect study conduct or the well-being of the subject
* History and/or presence of asthma or recurrent sinusitis. Active rhinitis at screening or upon admission to the study center.
* Any clinically significant nasal septum deviation, presence of septum perforations, and history of recurrent epistaxis and nasal polyps.
* Subjects with a history of sinus surgery and/or persistent hypertrophic inferior turbinates.
* History of vaccination with live vaccine within 7 days or attenuated vaccine within 14 days of the administration of the investigational product.
* Any clinically significant abnormalities in clinical laboratory safety assessment results
* A positive result at screening on serum hepatitis B surface antigen, hepatitis C antibodies and HIV antibodies.
* Significant orthostatic reaction at screening or upon admission to the study center as judged by the Principal Investigator.
* Abnormal vital signs, after 5 minutes supine rest,
* Any clinically significant abnormalities in rhythm, conduction, or morphology of resting electrocardiogram (ECG) that may interfere with the interpretation of QTc interval changes.
* Prolonged QTcF greater than 450 ms or shortened QTcF less than 360 ms or family history of long QT syndrome.
* Known or suspected drugs of abuse or alcohol abuse or dependence
* Positive screen for drugs of abuse or alcohol at screening or upon admission to the study center.
* Excessive intake of caffeine-containing foods or beverages within 48 hours prior to the admission to the study center.
* Use of drugs with enzyme-inducing properties such as St John's Wort, within 3 weeks prior to the administration of the investigational product.
* Abstain from smoking from 30 days prior to screening and for the duration of the study.
* Use of any prescribed medication as well as any over-the-counter/non prescribed/ herbal medicines, within 2 weeks prior to administration of the investigational product.
* Use of any nasal steroid 3 months prior to the administration of the investigational product.
* Involvement in the planning and/or conduct of the study
* Have received another new chemical entity or has participated in any other clinical study that included drug treatment within 3 months prior to administration of the investigational product in this study.
* Previous randomization of treatment in the present study or any other study with Flufirvitide-3.
* Plasma donation within 4 weeks prior to enrollment or blood donation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sam Hopkins, PhD, Study Director — Autoimmune Technologies, LLC
Locations (1):
- Quintiles Phase One Services, Overland Park, Kansas, United States